CLINICAL TRIAL: NCT03429439
Title: A Randomised Study on Intestinal Microbiota Transplantation for Chronic Hepatitis B Combined With Antiviral Therapy
Brief Title: Study on Effect of Intestinal Microbiota Transplantation in Chronic Hepatitis B
Acronym: CHB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017003
Record Dates: First submitted 2017-10-24; First posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2017-10

CONDITIONS: Chronic Hepatitis b
Keywords: chronic hepatitis B; intestinal microbiota transplantation; microbiota; antiviral therapy
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Fecal Microbiota Transplantation; Antiviral Agents

STUDY DESIGN:
Intervention Model Description: an open label, parallel study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMT Combined with Antiviral Therapy (Experimental): 60 chronic hepatitis B patients ongoing antiviral therapy will be recruited for the study, which involved a 6 times intestinal microbiota transplant and the time interval is generally 2 weeks.
  Interventions:
  Procedure: Intestinal Microbiota Transplantation Procedure: antiviral therapy
  Interventions: Other: intestinal microbiota transplant; Drug: Antiviral Agents
- Antiviral Agents (Other): 60 chronic hepatitis B patients ongoing antiviral therapy will be recruited for the study, which involved 12 months antiviral therapy.
  Interventions:
  Procedure: antiviral therapy
  Interventions: Drug: Antiviral Agents

INTERVENTIONS:
Other: intestinal microbiota transplant — Participants in experimental group take 6 times IMT with 2-week intervals.
  Arms: IMT Combined with Antiviral Therapy
Drug: Antiviral Agents — All participants continue present antiviral therapy over 12 months.

SUMMARY:
Chronic hepatitis B(CHB) is a common infectious disease affecting up to 2 billion people worldwide. Around 650 thousand people died of liver failure, cirrhosis and primary liver cancer caused by chronic hepatitis B every year. Age is the main factor affecting the chronicity of hepatitis B, while 90% and 25% to 30% of hepatitis b virus(HBV) infection in perinatal and infant period will develop into chronic infection respectively. Whereas the proportion in patients above 5 years old is only 5% to 10%. Intestinal microbiota plays an important role in maintaining normal physiological function of the intestine and the immune function of the body. It has been found that the disorder of intestinal microbiota is associated with numerous intestinal and parenteral diseases. Intestinal microbiota transplantation(IMT) is a significant method to reconstruct intestinal flora. Recently, the relationship between immune response and intestinal microbiota has been claimed. In a previous study using IMT to treat HBeAg positive chronic hepatitis B patients combined with antiviral therapy, 80% of them has reached HBeAg clearance. The investigators propose a randomised trial of IMT in patients with chronic hepatitis B combined with antiviral therapy. The investigators will assess the serum HBsAg, anti-HBs, HBeAg, anti-HBe, anti-hepatitis B core antigen, the relief of gastrointestinal symptoms, and the fecal microbiota before and after IMT. Patients will be randomized to either antiviral therapy or IMT combined antiviral therapy over a 26 weeks period.

DETAILED DESCRIPTION:
A group of 60 chronic hepatitis B patients combined with antiviral therapy will be recruited for study, which involved a 6 times IMT with gastroduodenoscopy and the time interval is generally 2 weeks. All participants will keep their present antiviral therapy. All participants will be assessed at baseline, after 1 months, 3 months, 6 months from baseline in order to evaluate the possible changes in:(1)Decrease of serum hepatitis B virus surface antigen(HBsAg) levels(as measured in IU/mL) and hepatitis B virus e antigen(HBeAg) levels(as measured in S/CO); (2)Appearance of serum anti-hepatitis B virus surface antigen(anti-HBs) and anti-hepatitis B virus e antigen(anti-HBe); (3)Relief of gastrointestinal symptoms:The onset and duration of gastrointestinal symptoms will be assessed by "Evaluation Score Table of Gastrointestinal Symptoms"; (4)Changes of gut microbiota: The changes of gut microbiota will be assessed by High-throughput sequencing (16S rRNA) in fecal samples from recruited patients before and after IMT.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent as appropriate
* 18 to 65 years of age
* No alcohol consumption or alcohol consumption <140g per week in men, and <70g per ween in women
* Been diagnosed with chronic hepatitis B

Exclusion Criteria:

* Alcoholic liver disease (ALD), chronic hepatitis C, autoimmune liver disease, Wilson's disease
* Drug treatment (tamoxifen, amiodarone, sodium valproate, methotrexate, glucocorticoids, etc.), total parenteral nutrition, inflammatory bowel disease, hypothyroidism, Cushing's syndrome, beta lipoprotein deficiency, insulin resistance related syndromes (lipid wasting diabetes mellitus, Mauriac syndrome), gastrointestinal surgery
* Hepatocellular carcinoma (HCC), biliary tract diseases and taking or taking chinese and western medicines that can lead liver enzymes elevation in the near future.
* Moderate and severe renal injury(serum creatinine>2mg/dL or 177mmol/L), moderate and severe chronic obstructive pulmonary disease, severe hypertension, cerebrovascular accident, congestive heart failure, unstable angina pectoris.
* Antibiotics treatment in 7 days before recruited and unwilling to stop it, long-term lipid-lowering drugs, antidiabetic drugs and other liver protecting drugs treatment
* Antibiotics, other probiotics, gastrointestinal motility drugs and other preparation that may influence intestinal microbiota treatment
* Other serious diseases that may interfere the recruitment or affect the survival, such as cancer or acquired immune deficiency syndrome
* Mentally or legally disabled person
* Preparing for pregnancy
* Medical or social condition which in the opinion of the principal investigator would interfere with or prevent regular follow up
* Participating in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-12-29 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Change of serum hepatitis B virus e antigen(HBeAg) level | 1 month, 3 months, 6months
  Serum hepatitis B virus e antigen(HBeAg) levels is measured in S/CO

SECONDARY OUTCOMES:
Change of serum hepatitis B virus surface antigen(HBsAg) level | 1 month, 3 months, 6months
  Serum hepatitis B virus surface antigen(HBsAg) levels is measured in IU/mL .
Change of serum anti-hepatitis B virus e antigen(anti-HBe) | 1 month, 3 months, 6months
  Appearance of serum anti-hepatitis B virus e antigen(anti-HBe) suggest the ability of body to resistant HBV.
Change of serum anti-hepatitis B virus surface antigen(anti-HBs) | 1 month, 3 months, 6months
  Appearance of serum anti-hepatitis B virus surface antigen(anti-HBs) suggest the ability of body to resistant HBV.
Changes of gut microbiota | 1 month, 3 months, 6months
  Alpha and Beta diversity of GI microbiota by High-throughput sequencing (16S rRNA) on baseline line and1 month, 3 months, 6months after treatment
relief of constipation | 1 month, 3 months, 6months
  The onset and duration of constipation will be assessed by "Evaluation Score Table of Gastrointestinal Symptoms".
relief of diarrhea | 1 month, 3 months, 6months
  The onset and duration of diarrhea will be assessed by "Evaluation Score Table of Gastrointestinal Symptoms".
relief of abdominal pain | 1 month, 3 months, 6months
  The onset and duration of abdominal pain will be assessed by "Evaluation Score Table of Gastrointestinal Symptoms".

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian, China

DOCUMENTS (2):
  • Study Protocol (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT03429439/Prot_000.pdf
  • Informed Consent Form (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT03429439/ICF_001.pdf